CLINICAL TRIAL: NCT03268798
Title: Unilateral Wrist Extension Training After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Dr. E. Paul Zehr, Professor, University of Victoria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D015017-2011-2015
Record Dates: First submitted 2017-08-24; First posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Stroke
Keywords: stroke; strength training; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Wrist extension training (Experimental)
  Interventions: Device: Unilateral wrist extension training

INTERVENTIONS:
Device: Unilateral wrist extension training — Participants will join a five-week training protocol with 3 sessions per week. During each session, 5 sets 5 maximal wrist extension training will be performed on participants less affected side.

SUMMARY:
Following stroke, muscle weakness and impaired motor function are expressed in both the more (MA; paretic) and less affected (LA; non-paretic) sides. Although the efficacy of resistance training is well recognized, training the MA limb directly may be initially difficult due to muscular weakness. "Cross-education" is training one side of the body increases strength in the untrained and opposite side. This concept can be applied in strength training when training the more affected sides cannot be initiated. Recently, our lab found six weeks of dorsiflexion resistance training in the LA leg improved the strength of both trained and untrained legs of chronic stroke participants.

The current project explored if cross-education exists in the upper limb in chronic stroke participants and if there are related changes in cortical and spinal cord plasticity. We hypothesized that unilateral strength in the less affected arm could enhance wrist extension strength bilaterally with related neural adoption and improved clinical function.

DETAILED DESCRIPTION:
Stroke produces muscle weakness seen on both more (paretic, MA) and less affected (non-paretic, LA) sides. "Cross-education" is training one side of the body increases strength or motor skill in the same muscles on the untrained side. This can be applied to enhance muscle strength in the MA side and we found that 6 weeks of dorsiflexion resistance training with the LA leg improved strength bilaterally in chronic stroke. To explore if cross-education occurs also in the upper limb after stroke, participants will complete a 5-week unilateral wrist extension training.

Twenty four participants will be recruited, 12 from Rehabilitation Neuroscience laboratory at University of Victoria, 12 from Brain Behaviour Laboratory at University of British Columbia. Before and after training, maximal voluntary contraction wrist extension force was measured with a 6-axis load cell using Cartesian coordinates (Fz = extension). Electromyography of extensor and flexor carpi radialis, biceps and triceps brachii were recorded. Fugl-Meyer and partial Wolf Motor Function Test were performed by the same physical therapist at each location. Reciprocal inhibition from wrist flexors to extensors, cutaneous reflexes evoked by median and superficial radial nerve stimulation were assessed in those at UVIC. Cortical silent period, short-interval intracortical inhibition, intracortical facilitation and transcallosal inhibition from transcranial magnetic stimulation were measured in participants at UBC.

ELIGIBILITY:
Inclusion Criteria:

* Over 6 months post-stroke;
* One side of arm shows muscle weakness
* Pass the screening test of Physical Activity Readiness Questionnaire
* Pass the screening test for dementia
* Free from dementia (score < 24 on the Montreal Cognitive Assessment) and any other contradiction for TMS test

Exclusion Criteria:

* Had medication affecting muscle tone within the past 3 months
* Wear a pacemaker

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-03; Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in wrist extension force | Week1-3: baselines were measured once per week for three times; Week 4-8: training(no measurement was taken); Week 9: post-test; Week 13: follow-up test
  To test if training could improve wrist extension strength, maximal wrist extension force were measured in both arms during the 3 baseline pretests, 1 post-test. There was a week in between each baseline tests, post-test will be performed within one week after the training finished. To test if the force changes maintained after training, follow-up test was performed 5 weeks after training finished.

SECONDARY OUTCOMES:
Changes in the modulation of spinal-mediated muscle reflexes | Week1-3: baselines were measured once per week for three times; Week 4-8: training(no measurement was taken); Week 9: post-test;
  To test if training could induce neural adaptation at spinal level, spinal-mediated muscle reflexes include reciprocal inhibition and cutaneous reflexes in the wrist extensor muscle were measured. Muscle reflex amplitudes were compared before and after training. There was no follow-up test for this measurement
Neural adaptation in the corticospinal pathway | Week1-3: baselines were measured once per week for three times; Week 4-8: training(no measurement was taken); Week 9: post-test;
  To test if training could induced neural adaptation at corticospinal level, cortical silent period, short-interval intracortical inhibition, intracortical facilitation and transcallosal from transcranial magnetic stimulation were measured in wrist extensor muscle. Changes in the muscle reflex amplitudes and cortical silent period duration were compared before and after training. There was no follow-up test for this measurement.
Upper limb impairment assessments | Week1-3: baselines were measured once per week for three times; Week 4-8: training(no measurement was taken); Week 9: post-test;
  Fugl-Meyer test score were assessed by licensed physiotherapists. Scores were compared before and after training. There was no follow-up test for this measurement.
Upper limb function assessments | Week1-3: baselines were measured once per week for three times; Week 4-8: training (no measurement was taken); Week 9: post-test; Week 13: follow-up test
  Wolf Motor Function Test were assessed by licensed physiotherapists. Scores were compared before and after training.
Ten-meter walking test | Week1-3: baselines were measured once per week for three times; Week 4-8: training (no measurement was taken); Week 9: post-test;
  Walking speed was compared before and after training. There was no follow-up test for this measurement
Six-minute walking test | Week1-3: baselines were measured once per week for three times; Week 4-8: training(no measurement was taken); Week 9: post-test;
  Walking distance was compared before and after training. There was no follow-up test for this measurement
Timed up and go | Week1-3: baselines were measured once per week for three times; Week 4-8: training(no measurement was taken); Week 9: post-test;
  Walking speed was compared before and after training. There was no follow-up test for this measurement.

CONTACTS AND LOCATIONS:
Overall Officials: E.Paul Zehr, Principal Investigator — Rehabilitation Neuroscience Laboratory, University of Victoria